CLINICAL TRIAL: NCT03705715
Title: Identifying Correlates of Brain Microglial Activation in Neuropsychiatric Syndromes: a Dimensional Approach
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Alan Prossin, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-15-0744
Record Dates: First submitted 2015-12-10; First posted 2018-10-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Neuropsychiatric Syndromes
Keywords: Microglial activation; Immune activation; PET neuroimaging
MeSH Terms: interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PET with radiotracer [11C]PBR-28 or [11C]ER176 (Experimental): PET with radiotracer [11C]PBR-28 or [11C]ER176 will be performed. [11C]PBR-28 or [11C]ER176 will be injected into subjects' veins during PET scanning.
  Interventions: Drug: PET with radiotracer [11C]PBR-28 ( or [11C]ER176)
- PET with radiotracer [11C]PBR-28 or [11C]ER176 and affective challenge (Experimental): PET with radiotracer [11C]PBR-28 or [11C]ER176 will be performed. [11C]PBR-28 or [11C]ER176 will be injected into subjects' veins during PET scanning. Affective challenge (e.g. induction of mood, affective pain) will be presented to the patient during the PET scanning period.

INTERVENTIONS:
Drug: PET with radiotracer [11C]PBR-28 ( or [11C]ER176) — [11C]PBR-28 or [11C]ER176 will be injected into subjects' veins during PET scanning.
  Other Names: [O-methyl-11C]N-acetyl-N-(2-methoxybenzyl)-2-phenoxy- 5-pyridinamine
  Arms: PET with radiotracer [11C]PBR-28 or [11C]ER176
Other: Affective challenge — Affective challenge is the induction of, for example, mood or affective pain.
  Other Names: biobehavioral challenges

SUMMARY:
The purpose of this research is to determine whether there is more extensive inflammation in the brain of people with clinical evidence of neuropsychiatric syndromes, such as mood disorder, chronic pain syndrome, dementia, traumatic brain injury, or substance abuse. The research will also explore whether there is more inflammation in patients with more neuropsychiatric symptoms. Inflammation in the brain will identified by using Positron Emission Tomography (PET) with the radiotracer [11C]PBR-28 or [11C]ER176.

DETAILED DESCRIPTION:
This study will explore whether brain microglial activation (which leads to an inflammatory response) is more extensive in individuals with clinical evidence of neuropsychiatric syndromes and whether the extent of microglial activation is proportional to the extent of neuropsychiatric symptoms.

More specifically, the hypothesis is that:

1. Brain microglial activation is more substantial in the presence of neuropsychiatric illness, and the extent of brain microglial activation is proportional to severity of phenotypic presentation of neuropsychiatric illness (i.e. depression, cognitive impairment, fatigue, etc.) in a given patient.
2. Specific brain regions where enhanced microglial activation is present underlie a portion of phenotypic variance in neuropsychiatric patients
3. Combinations of neuropsychiatric phenotypes rather than specific differences in immune mechanisms underlie the contribution of central immune activation to a specific neuropsychiatric diagnosis.

The following measures will be obtained:

1. microglial activation as quantified by PET using the radiotracer [11C]PBR-28 or [11C]ER176. ([11C]PBR-28 and [11C]ER176 specifically bind translocator protein (TSPO), which is associated with microglial activation and can thus serve as an in vivo biomarker of microglial activation and neuroinflammation. TSPO is also called the peripheral benzodiazepine receptor (PBR))
2. dimension of specific neuropsychiatric symptoms (Hamilton Depression Rating Scale (HDRS), Montreal Cognitive Assessment (MoCA), Positive and Negative Affect Schedule (PANAS))
3. presence/absence of a specific neuropsychiatric diagnosis (Dementing Illnesses, Traumatic Brain Injury, Major Depression, Bipolar Disorder, Pain Syndromes, Other Affective Disorders, etc.)

Using the above measures, correlations (and brain regional correlations) between the extent of microglial activation and the presence of a dimension of neuropsychiatric symptoms will be tested for. Following this, the presence of microglial activation (and brain regional microglial activation) 1) between healthy control volunteers and volunteers with neuropsychiatric syndromes and 2) between the various neuropsychiatric syndromes/diagnoses will be tested for.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-80 years old
* Males or females
* Must be right handed
* Must be able to sit unaccompanied for long periods of time with little body movement
* Must be illicit drug free at time of scanning as appropriate (UDS negative),
* Must be either healthy (without medical, neurological, psychiatric illness) or have a diagnosis of a neuropsychiatric syndrome (mood disorder, chronic pain syndrome, dementias, traumatic brain injury, substance/alcohol use disorder).
* Healthy Control volunteers must be medication free (≥ 14 days)
* Illicit drug free at time of scanning (verified by negative urine drug screen)

Exclusion Criteria:

* Must not be a smoker.
* Females must not be pregnant or nursing.
* Must not suffer from claustrophobia
* Must not meet exclusion criteria for MRI scanning (i.e. non-fixed magnetisable objects)
* Must not be PBR-28 low affinity binder (or using the [11C]ER176 study radiotracer)
* Healthy control volunteers must not have on-going, chronic, or relapsing/remitting medical, psychiatric (absence of both DSM-IV Axis I and/or Axis II disorders), or neurological illness as determined by combination of history, medical record, and/or examination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Level of TSPO expression as quantified by PET imaging to detect binding of the TSPO radiotracer [11C]PBR-28 | obtained during PET scanning (between 1:30 PM and 3 PM) at study baseline within a few days of study enrollment

SECONDARY OUTCOMES:
Affect as measured by the Hamilton Depression Rating Scale (HDRS) | within 1-2 hours before PETobtained during PET scanning (between 1:30 PM and 3 PM) at study baseline within a few days of study enrollment
  HDRS is a multiple item questionnaire used to provide an indication of depression. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression.
Mental Status as measured by the Montreal Cognitive Assessment (MoCA) | within 1-2 hours before PETobtained during PET scanning (between 1:30 PM and 3 PM) at study baseline within a few days of study enrollment
  The MoCA assesses several cognitive domains. The total possible score is 30 points with a score of 26 or more considered normal.
Affect as measured by the Positive and Negative Affect Schedule (PANAS) | within 1-2 hours before PETobtained during PET scanning (between 1:30 PM and 3 PM) at study baseline within a few days of study enrollment
  Positive Affect Score: Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score: Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Affect as measured by the Positive and Negative Affect Schedule (PANAS) | during PET (between 1:30 PM and 3 PM)obtained during PET scanning (between 1:30 PM and 3 PM) at study baseline within a few days of study enrollment
  Positive Affect Score: Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score: Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.
Affect as measured by the Positive and Negative Affect Schedule (PANAS) | immediately following PET (3PM +/- 30 minutes)obtained during PET scanning (between 1:30 PM and 3 PM) at study baseline within a few days of study enrollment
  Positive Affect Score: Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. Negative Affect Score: Scores can range from 10 - 50, with lower scores representing lower levels of negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Prossin, MBBS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- BBSB at UTHealth, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No